CLINICAL TRIAL: NCT02365337
Title: Influence of Serum Vitamin D Levels on Embryo Morphokinetic Parameters in Women Undergoing Controlled Ovarian Hyperstimulation
Brief Title: Influence of Serum Vitamin D Levels on Embryo Morphokinetic Parameters
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bahceci Clinic (Other)
Responsible Party: Principal Investigator, C CELİK, Associate Professor, Bahceci Clinic
Other Study IDs: BHC19771981
Record Dates: First submitted 2015-02-09; First posted 2015-02-18 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Infertility
Keywords: Vitamin D; time lapse monitoring; embryo
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- vitamin D levels < 20ng/ ml: Vitamin D levels < 20ng/ ml
- vitamin D levels>20ng/ ml: Vitamin D levels >20ng/ ml

SUMMARY:
The aim of this study is observing the relation between serum Vitamin D levels and morphokinesis of time lapse monitored Day 5 embryo in between 18 and 38 years age women undergoing controlled ovarian hyperstimulation (COH) because of unexplained or tubal factor infertility. Individuals will be divided into 2 groups according to serum vitamin D levels as normal or low , and the influence of those levels in morphokinetic parameters of embryos will be identified.

DETAILED DESCRIPTION:
Up to date there are few studies questioning the serum Vitamin D deficiency as a negative factor for pregnancy rates in women undergoing COH cycles and also are displaying different and inconclusive results. This dedicated negative affects may be mediated through endometrial and/or ovarial factors. In experimental animal models Vitamin D receptors have been found in endometrium and ovaries and deficient levels might have been a cause of impaired folliculogenesis. In one of human study Vitamin D has been suggested as a positive regulator of anti- Mullerian hormone (AMH) production. Therefore, we aimed to clarify the affects of Vitamin D on folliculogenesis, oogenesis and embryo quality in COH cycles by using time lapse monitoring.

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 38 years age, 2 or less in vitro fertilization (IVF) / intracytoplasmic sperm injection (ICSI) attempt history, Unexplained or tubal factor infertility, Serum Follicle Stimulating Hormone (FSH) < 10, Antral Follicule Count (AFC)> 6-8

Exclusion Criteria:

* Male factor infertility, Presence of endometriosis or adenomyosis,Diminished ovarian reserve

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: participants will be recruited among infertile women who is seeking for IVF treatment and fullfilling the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-06 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
time to 2 pronucleus (PN) membrane breakdown, first cleavage and 3, 4, 5, 6, 7, and 8 cells stages, morula and blastocyst stage (t2, t3, t4, t5, t6, t7, t8, t Morula (M), t Blastocyst (B) ) | between 17 and 120 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Bahceci Fulya IVF Center, Istanbul, Fulya, Turkey (Türkiye)

REFERENCES:
- [Background] Dennis NA, Houghton LA, Jones GT, van Rij AM, Morgan K, McLennan IS. The level of serum anti-Mullerian hormone correlates with vitamin D status in men and women but not in boys. J Clin Endocrinol Metab. 2012 Jul;97(7):2450-5. doi: 10.1210/jc.2012-1213. Epub 2012 Apr 16. PMID 22508713